CLINICAL TRIAL: NCT03156959
Title: Efficacy of Eye Movement Desensitization and Reprocessing (EMDR) Plus Broad Form of Enhanced Cognitive Behavioural Therapy (CBT-Eb) in Patients With Eating Disorders. A Randomized Controlled Trial
Brief Title: CBT-Eb Plus EMDR Versus CBT-Eb in Patients With Eating Disorders
Acronym: TREAT-EMDR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruggeri, Mirella (Other)
Responsible Party: Sponsor-Investigator, Ruggeri, Mirella, Full Professor in Psychiatry, Universita di Verona
Organization: Universita di Verona (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1153CESC
Record Dates: First submitted 2017-05-08; First posted 2017-05-17 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Eating Disorder
Keywords: Eating disorders; Cognitive Behavioral Therapy; Eye Movement Desensitization and Processing
MeSH Terms: conditions — Feeding and Eating Disorders | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMDR plus CBT-Eb (Experimental): 20 CBT-Eb sessions will be mandatory for patients with BMI>17.5 and 40 CBT-Eb sessions will be mandatory for patients with BMI≤17.5. In the EMDR plus CBT-Eb arm, 16 EMDR sessions will be mandatory in adjunction to the CBT-Eb sessions, irrespectively of the BMI. EMDR will use an eight-phase approach that will include having the patient recall distressing images while receiving one of several types of bilateral sensory input, such as side to side eye movements.
  Patients will follow psychopharmacological treatment for anxiety and depression symptoms if needed, and their parents will be invited to participate to a cycle of eight family meetings on eating disorders and psychological support following ECHO approach (Rhind et al., 2014).
  Interventions: Behavioral: EMDR; Behavioral: CBT-Eb
- CBT-Eb alone (Active Comparator): 20 CBT-Eb sessions will be mandatory for patients with BMI>17.5 and 40 CBT-Eb sessions will be mandatory for patients with BMI≤17.5.
  Patients will follow psychopharmacological treatment for anxiety and depression symptoms if needed, and their parents will be invited to participate to a cycle of eight family meetings on eating disorders and psychological support following ECHO approach (Rhind et al., 2014).
  Interventions: Behavioral: CBT-Eb

INTERVENTIONS:
Behavioral: EMDR — The Eye Movement Desensitization and Reprocessing (EMDR) is a psychotherapy developed by Francine Shapiro (2001) that emphasizes disturbing memories as the cause of psychopathology. These memories and associated stimuli are inadequately processed and stored in an isolated memory network (Shapiro and Laliotis, 2010). The goal of EMDR is to reduce the long-lasting effects of distressing memories by developing more adaptive coping mechanisms.
  Arms: EMDR plus CBT-Eb
Behavioral: CBT-Eb — The broad form of Enhanced Cognitive Behavioural Therapy (CBT-Eb; Fairburn and colleagues, 2009) addresses psychopathological processes "external" to the eating disorder, such as clinical perfectionism, low self-esteem or interpersonal difficulties, which interact with the disorder itself.

SUMMARY:
Enhanced CBT (CBT-E) is an effective treatment for the majority of outpatients with an eating disorder; however in about 30% of patients remission is made difficult. This may be due to the concomitant presence of trauma. Therefore we expect that a combination of CBT-E and EMDR, which is the evidence based treatment for PTSD disorder, would enhance the remission probability. This trial has a parallel group randomized controlled design. All patients who will enter in contact with the Regional Reference Centre for Eating Disorders in Verona and will satisfy inclusion criteria will be randomized to the broad form of CBT-E (CBT-Eb) plus EMDR or CBT-Eb alone. Patients will be evaluated before the treatment, at the end of treatment and after 6 months post-treatment with a set of standardized measure to assess eating disorder symptoms and other possible predisposing and moderating factors. The efficacy of CBT-E vs CBT-E + EMDR will be evaluated at the end of the treatment and after 6 months in terms of global score of the Eating Disorder Examination. Moreover the changes in other secondary outcomes will be considered. This explorative study may suggest new hypothesis for larger RCTs in order to increase the knowledge on ED.

DETAILED DESCRIPTION:
Background. The Diagnostic and Statistical Manual of Mental Disorders fifth edition (DSM-5) distinguishes three broad categories of Eating Disorder (ED): anorexia nervosa (AN), bulimia nervosa (BN), and Other Specified Feeding or Eating Disorder (OSFED). The International Classification of Diseases tenth revision (ICD-10) also reports three categories: anorexia nervosa, bulimia nervosa, and atypical eating disorder.

Anorexia Nervosa (AN). Anorexia nervosa, which primarily affects adolescent girls and young women, is characterized by distorted body image and excessive dieting that lead to severe weight loss with a pathological fear of becoming fat. People affected by anorexia often go to great attempts to hide their behaviour from family and friends. Often people with anorexia have low confidence and poor self-esteem. They can see their weight loss as a positive achievement that can help increase their confidence. It can also contribute to a feeling of gaining control over body weight and shape. The illness can affect people's relationship with family and friends, causing them to withdraw; it can also have an impact on how they perform in education or at work. The seriousness of the physical and emotional consequences of the condition is often not acknowledged or recognised and people with anorexia often do not seek help.

Bulimia Nervosa (BN). Bulimia nervosa is a serious disorder that involves a recurring pattern of binge eating followed by dangerous compensatory behaviours in an effort to counteract or "undo" the calories consumed during the binge. Marked distress regarding binge eating is present. The binge eating occurs, on average, at least once a week for three months. People with bulimia often feel trapped in this cycle of dysregulated eating, and there is a risk for major medical consequences associated with bulimic behaviours.

Other Specified Feeding or Eating Disorder (OSFED). It is a feeding or eating disorder that causes significant distress or impairment, but does not meet the criteria for another feeding or eating disorder.

Treatment of Eating Disorders. Guidelines recommended that people with anorexia nervosa should first be offered outpatient treatment and that inpatient care be used for those who do not respond or who present with high risk and little psychosocial resources. Nevertheless the evidence base relating to the treatment of anorexia nervosa is meagre and no first line treatment is identified. Recommendations emphasise the importance of a multi-disciplinary approach including medical, nutritional, social, and psychological components. Among psychotherapies, CBT is one of the suggested treatment. For atypical eating disorders (eating disorders not otherwise specified), in the absence of evidence "it is recommended that the clinician considers following the guidance on the treatment of the eating problem that most closely resembles the individual patient's eating disorder". Regarding bulimia nervosa, CBT-BN is recommended as first-line treatment. CBT-BN has evolved over the past decade in response to a variety of challenges: its procedures have been refined, particularly those addressing patients over evaluation of shape and weight, and it has been adapted to make it suitable for all forms of eating disorder, thereby making it "transdiagnostic" in its scope. This implemented CBT treatment was defined Enhanced CBT. Several studies addressed the efficacy of CBT-E across several eating disorders. In detail, there are two possible CBT treatments for eating disorders, a simpler one, more focused on eating disorders features defined as focused form of Enhanced CBT (CBT-Ef) and another more complex, that addresses external psychopathological processes, named broad form of Enhanced CBT (CBT-Eb). This new version of the treatment also addresses psychopathological processes "external" to the eating disorder, such as clinical perfectionism, low self-esteem or interpersonal difficulties, which interact with the disorder itself.

Eating Disorders and Trauma History. There is evidence of an association among multiple episodes or forms of trauma, ED and the level of post-traumatic symptoms. Many studies have documented trauma history in patients with ED, with childhood sexual abuse being the most well-documented trauma in these patients. Other types of trauma reported in ED patients include physical and emotional abuse, teasing and bullying, and parental break-up and loss of a family member. A review emphasized that trauma histories are much more commonly associated with BN, AN binge-purge type, and EDNOS characterized by bulimic symptoms, such as binge eating disorder (BED) or "purging disorder," than with AN restricting type or EDNOS not associated with bulimic symptoms. Bulimic women had more psychopathology than non-bulimic women, and there is an association between the severity of comorbid psychopathology and the severity of trauma. It has been suggested that it is PTSD, rather than an abuse history per se, that best forecasts the emergence of BN. In addition, PTSD predicts comorbidity with major depression and alcohol abuse/substance dependence in conjunction with BN. PTSD prevalence in ED patients is about 24.3%, confirming the comorbidity between both disorders. It has been suggested that there is no significant difference between AN and BN patients with regard to the lifetime prevalence of trauma. Some authors underline that patients with higher PTSD symptomatology also suffer from more severe ED symptoms. As far as regards PTSD treatment, CBT with prolonged exposure, eye movement desensitization and reprocessing (EMDR), and pharmacotherapy have shown to be the most effective. EMDR is a psychotherapy that emphasizes disturbing memories as the cause of psychopathology. These memories and associated stimuli are inadequately processed and stored in an isolated memory network. The goal of EMDR is to reduce the long-lasting effects of distressing memories by developing more adaptive coping mechanisms. The therapy uses an eight-phase approach that includes having the patient recall distressing images while receiving one of several types of bilateral sensory input, such as side to side eye movements. The use of pharmacotherapy without concomitant psychotherapy is generally ineffective in terms of producing complete and lasting abstinence in ED patients. It is important to assess the mechanisms that functionally link disorders or problem behaviours together. This is particularly true for those with PTSD and other trauma-related comorbidity. In this respect, EMDR appears to easily complement the CBT for PTSD. EMDR has been shown to be as efficacious as CBT with prolonged exposure as well as treatment with fluoxetine. There are also some clinical reports which support the adoption of EMDR to treat ED.

Aim. The trial described here has the aim to compare, at the end of the treatment and at 6 months post-treatment, the efficacy of Eye Movement Desensitization and Reprocessing (EMDR) plus Broad Form of Enhanced Cognitive Behavioural Therapy (CBT-Eb) with that of Broad Form of Cognitive-Behavioural Therapy (CBT-Eb) alone in a sample of patients with Eating Disorders. We expect that EMDR plus CBT-Eb will ameliorate the severity of the eating disorder compared to CBT-Eb alone, primarily in patients with trauma history.

Design. The trial has a parallel group randomized controlled design, which compares, at the end of the treatment and after 6 months post-treatment, the efficacy of Eye Movement Desensitization and Reprocessing (EMDR) plus Broad Form of Enhanced Cognitive Behavioural Therapy (CBT-Eb) with that of Broad Form of Cognitive-Behavioural Therapy (CBT-Eb) alone in a sample of patients with Eating Disorders.

Participants. Study participants are recruited from the Regional Reference Centre for Eating Disorders operating for the Italian National Health Service in Verona. Those who satisfy inclusion and exclusion criteria and give written informed consent to participate in the study will be randomized to CBT-Eb plus EMDR or CBT-Eb alone.

Clinical assessment. At baseline, at the conclusion of the treatment and at 6 months post-treatment, patients will be assessed by the following set of standardized instruments:

* Eating Disorder Examination (EDE)
* Hopkins Symptom Checklist (SCL-90)
* Eating Disorders Inventory (EDI.3)
* Barratt Impulsiveness Scale (BIS-11)
* Level of Expressed Emotion (LEE)
* Young Schema Questionnaire (YSQ)
* Penn State Worry Questionnaire (PSWQ)
* Rathus Assertiveness Scale (RAS)
* Clinical Impairment Assessment Questionnaire (CIA)
* Semi-structured Interview for Eating Disorder (ISDA)
* Parental Bonding Instrument (PBI)
* Childhood Experience of Care and Abuse Questionnaire (CECA-Q)
* Family History Screen
* Tridimensional Personality Questionnaire (TPQ)
* Impact of Event Scale - Revised (IES-R)
* Inventario degli Eventi Stressanti e Traumatici della Vita
* Global Assessment of Functioning (GAF)
* Dissociative Experience Scale (DIS-Q)
* Toronto Alexithymia Scale (TAS-20)
* Hypomania/Mania Symptom Checklist (HCL-32)
* Scheda ad hoc sugli interventi ricevuti. Randomization procedure. 40 patients will be allocated to CBT-Eb plus EMDR treatment and 40 patients to CBT-Eb treatment alone. Patients will be randomly assigned to one of the two trial arms with a 1:1 allocation rate. Stratified randomization will be performed to balance differences in patients' characteristics [trauma (yes vs no) and BMI (<=17.5 vs >17.5)].

Sample size and power calculations. A total of 80 patients (40 patients per treatment condition) will detect a difference in terms of global EDE score of 0.64, with a power of 80% (two-side t test at 0.05), assuming a standard deviation of global EDE score of 1.0. The sample size has been estimated by using PASS 11.

Statistical analysis. Statistical analysis will be based on an intention-to-treat (ITT) basis, comparing outcomes from all patients allocated to the two trial arms. The ITT principle will allow for potential biases arising from loss to follow-up, under the assumption that missing outcomes are missing at random (MAR). Findings will be reported according to the CONSORT guidelines for parallel group randomised trials.

ELIGIBILITY:
Inclusion Criteria:

* Age between 14 and 45 years
* Diagnosis of Eating Disorder that meets DSM 5 diagnostic criteria for Anorexia Nervosa (AN), Bulimia Nervosa (BN) or Other Specified Feeding or Eating Disorder (OSFED)
* A clinical severity which permits to treat the person at out-patient level

Exclusion Criteria:

* Eating Disorder of high clinical severity, not treatable at out-patient level
* Comorbidity with psychotic symptoms or any other DSM 5 disorder which might hinder eating disorder treatment
* Medical conditions which might impede data interpretation (chemotherapy, pregnancy status)
* Substances use and abuse
* Having previously received an evidence-based CBT treatment for the same eating disorder and/or EMDR

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-06-19 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Severity of the Eating Disorder | From BL to t1 (at 9 months if BMI>17.5 and 14 months if BMI<=17.5)
  Global score of the Eating Disorder Examination (EDE)
Changes in Severity of the Eating Disorder | From t1 (at 9 months from BL if BMI>17.5 and 14 months from BL if BMI<=17.5) to t2 (after 6 months from t1)
  Global score of the Eating Disorder Examination (EDE)

SECONDARY OUTCOMES:
Changes in Psychopathological conditions | From BL to t1 (at 9 months if BMI>17.5 and 14 months if BMI<=17.5)
  Hopkins Symptom Checklist (SCL-90)
Changes in Psychopathological conditions | From t1 (at 9 months from BL if BMI>17.5 and 14 months from BL if BMI<=17.5) to t2 (after 6 months from t1)
  Hopkins Symptom Checklist (SCL-90)
Changes in the Number of patients "in remission" for general psychopathology | From BL to t1 (at 9 months if BMI>17.5 and 14 months if BMI<=17.5)
  Global SCL-90 score less than 1
Changes in the Number of patients "in remission" for general psychopathology | From t1 (at 9 months from BL if BMI>17.5 and 14 months from BL if BMI<=17.5) to t2 (after 6 months from t1)
  Global SCL-90 score less than 1
Changes in Eating disorder risk factors | From BL to t1 (at 9 months if BMI>17.5 and 14 months if BMI<=17.5)
  Eating Disorders Inventory (EDI.3)
Changes in Eating disorder risk factors | From t1 (at 9 months from BL if BMI>17.5 and 14 months from BL if BMI<=17.5) to t2 (after 6 months from t1)
  Eating Disorders Inventory (EDI.3)
Changes in Subjective impact of traumatic events | From BL to t1 (at 9 months if BMI>17.5 and 14 months if BMI<=17.5)
  Impact of Event Scale-Revised (IES-R)
Changes in Subjective impact of traumatic events | From t1 (at 9 months from BL if BMI>17.5 and 14 months from BL if BMI<=17.5) to t2 (after 6 months from t1)
  Impact of Event Scale-Revised (IES-R)
Changes in Intensity of dissociative experiences | From BL to t1 (at 9 months if BMI>17.5 and 14 months if BMI<=17.5)
  Dissociative Experience Scale (DIS-Q)
Changes in Intensity of dissociative experiences | From t1 (at 9 months from BL if BMI>17.5 and 14 months from BL if BMI<=17.5) to t2 (after 6 months from t1)
  Dissociative Experience Scale (DIS-Q)
Changes in Caregiver expressed emotions (from the patient point of view) | From BL to t1 (at 9 months if BMI>17.5 and 14 months if BMI<=17.5)
  Level of Expressed Emotions (LEE)
Changes in Caregiver expressed emotions (from the patient point of view) | From t1 (at 9 months from BL if BMI>17.5 and 14 months from BL if BMI<=17.5) to t2 (after 6 months from t1)
  Level of Expressed Emotions (LEE)
Changes in Global functioning | From BL to t1 (at 9 months if BMI>17.5 and 14 months if BMI<=17.5)
  Global Assessment of Functioning (GAF)
Changes in Global functioning | From t1 (at 9 months from BL if BMI>17.5 and 14 months from BL if BMI<=17.5) to t2 (after 6 months from t1)
  Global Assessment of Functioning (GAF)
Changes in Level of impulsiveness | From BL to t1 (at 9 months if BMI>17.5 and 14 months if BMI<=17.5)
  Barratt Impulsiveness Scale (BIS-11)
Changes in Level of impulsiveness | From t1 (at 9 months from BL if BMI>17.5 and 14 months from BL if BMI<=17.5) to t2 (after 6 months from t1)
  Barratt Impulsiveness Scale (BIS-11)
Changes in Alexithymia | From BL to t1 (at 9 months if BMI>17.5 and 14 months if BMI<=17.5)
  Toronto Alexithymia Scale (TAS-20)
Changes in Alexithymia | From t1 (at 9 months from BL if BMI>17.5 and 14 months from BL if BMI<=17.5) to t2 (after 6 months from t1)
  Toronto Alexithymia Scale (TAS-20)
Changes in Assertiveness | From BL to t1 (at 9 months if BMI>17.5 and 14 months if BMI<=17.5)
  Rathus Assertiveness Scale (RAS)
Changes in Assertiveness | From t1 (at 9 months from BL if BMI>17.5 and 14 months from BL if BMI<=17.5) to t2 (after 6 months from t1)
  Rathus Assertiveness Scale (RAS)
Changes in Brooding | From BL to t1 (at 9 months if BMI>17.5 and 14 months if BMI<=17.5)
  Penn State Worry Questionnaire (PSWQ)
Changes in Brooding | From t1 (at 9 months from BL if BMI>17.5 and 14 months from BL if BMI<=17.5) to t2 (after 6 months from t1)
  Penn State Worry Questionnaire (PSWQ)
Changes in Psychosocial damage | From BL to t1 (at 9 months if BMI>17.5 and 14 months if BMI<=17.5)
  Clinical Impairment Assessment Questionnaire (CIA)
Changes in Psychosocial damage | From t1 (at 9 months from BL if BMI>17.5 and 14 months from BL if BMI<=17.5) to t2 (after 6 months from t1)
  Clinical Impairment Assessment Questionnaire (CIA)
Changes in Hypomanic or manic symptoms | From BL to t1 (at 9 months if BMI>17.5 and 14 months if BMI<=17.5)
  Hypomania/Mania Symptom Checklist (HCL-32)
Changes in Hypomanic or manic symptoms | From t1 (at 9 months from BL if BMI>17.5 and 14 months from BL if BMI<=17.5) to t2 (after 6 months from t1)
  Hypomania/Mania Symptom Checklist (HCL-32)
Changes in Maladaptive schemes | From BL to t1 (at 9 months if BMI>17.5 and 14 months if BMI<=17.5)
  Young Schema Questionnaire (YSQ)
Changes in Maladaptive schemes | From t1 (at 9 months from BL if BMI>17.5 and 14 months from BL if BMI<=17.5) to t2 (after 6 months from t1)
  Young Schema Questionnaire (YSQ)

CONTACTS AND LOCATIONS:
Overall Officials: Mirella Ruggeri, Prof, Study Chair — University of Verona, Section of Psychiatry
Locations (1):
- Regional Reference Centre For Eating Disorders of Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brewerton TD. Eating disorders, trauma, and comorbidity: focus on PTSD. Eat Disord. 2007 Jul-Sep;15(4):285-304. doi: 10.1080/10640260701454311. PMID 17710567
- [Background] Dansky BS, Brewerton TD, Kilpatrick DG, O'Neil PM. The National Women's Study: relationship of victimization and posttraumatic stress disorder to bulimia nervosa. Int J Eat Disord. 1997 Apr;21(3):213-28. doi: 10.1002/(sici)1098-108x(199704)21:33.0.co;2-n. PMID 9097195
- [Background] Murphy R, Straebler S, Cooper Z, Fairburn CG. Cognitive behavioral therapy for eating disorders. Psychiatr Clin North Am. 2010 Sep;33(3):611-27. doi: 10.1016/j.psc.2010.04.004. PMID 20599136
- [Background] Fairburn CG, Jones R, Peveler RC, Hope RA, O'Connor M. Psychotherapy and bulimia nervosa. Longer-term effects of interpersonal psychotherapy, behavior therapy, and cognitive behavior therapy. Arch Gen Psychiatry. 1993 Jun;50(6):419-28. doi: 10.1001/archpsyc.1993.01820180009001. PMID 8498876
- [Background] Fairburn CG, Bailey-Straebler S, Basden S, Doll HA, Jones R, Murphy R, O'Connor ME, Cooper Z. A transdiagnostic comparison of enhanced cognitive behaviour therapy (CBT-E) and interpersonal psychotherapy in the treatment of eating disorders. Behav Res Ther. 2015 Jul;70:64-71. doi: 10.1016/j.brat.2015.04.010. Epub 2015 Apr 22. PMID 26000757
- [Background] Fairburn CG, Cooper Z, Doll HA, O'Connor ME, Bohn K, Hawker DM, Wales JA, Palmer RL. Transdiagnostic cognitive-behavioral therapy for patients with eating disorders: a two-site trial with 60-week follow-up. Am J Psychiatry. 2009 Mar;166(3):311-9. doi: 10.1176/appi.ajp.2008.08040608. Epub 2008 Dec 15. PMID 19074978
- [Background] Foa EB, Dancu CV, Hembree EA, Jaycox LH, Meadows EA, Street GP. A comparison of exposure therapy, stress inoculation training, and their combination for reducing posttraumatic stress disorder in female assault victims. J Consult Clin Psychol. 1999 Apr;67(2):194-200. doi: 10.1037//0022-006x.67.2.194. PMID 10224729
- [Background] Follette VM, Polusny MA, Bechtle AE, Naugle AE. Cumulative trauma: the impact of child sexual abuse, adult sexual assault, and spouse abuse. J Trauma Stress. 1996 Jan;9(1):25-35. doi: 10.1007/BF02116831. PMID 8750449
- [Background] Grilo CM, Masheb RM. Childhood maltreatment and personality disorders in adult patients with binge eating disorder. Acta Psychiatr Scand. 2002 Sep;106(3):183-8. doi: 10.1034/j.1600-0447.2002.02303.x. PMID 12197855
- [Background] Kent A, Waller G, Dagnan D. A greater role of emotional than physical or sexual abuse in predicting disordered eating attitudes: the role of mediating variables. Int J Eat Disord. 1999 Mar;25(2):159-67. doi: 10.1002/(sici)1098-108x(199903)25:23.0.co;2-f. PMID 10065393
- [Background] Mahon J, Bradley SN, Harvey PK, Winston AP, Palmer RL. Childhood trauma has dose-effect relationship with dropping out from psychotherapeutic treatment for bulimia nervosa: a replication. Int J Eat Disord. 2001 Sep;30(2):138-48. doi: 10.1002/eat.1066. PMID 11449447
- [Background] Reyes-Rodriguez ML, Von Holle A, Ulman TF, Thornton LM, Klump KL, Brandt H, Crawford S, Fichter MM, Halmi KA, Huber T, Johnson C, Jones I, Kaplan AS, Mitchell JE, Strober M, Treasure J, Woodside DB, Berrettini WH, Kaye WH, Bulik CM. Posttraumatic stress disorder in anorexia nervosa. Psychosom Med. 2011 Jul-Aug;73(6):491-7. doi: 10.1097/PSY.0b013e31822232bb. Epub 2011 Jun 28. PMID 21715295
- [Background] Rorty M, Yager J, Rossotto E. Childhood sexual, physical, and psychological abuse and their relationship to comorbid psychopathology in bulimia nervosa. Int J Eat Disord. 1994 Dec;16(4):317-34. doi: 10.1002/1098-108x(199412)16:43.0.co;2-j. PMID 7866412
- [Background] Rothbaum BO, Astin MC, Marsteller F. Prolonged Exposure versus Eye Movement Desensitization and Reprocessing (EMDR) for PTSD rape victims. J Trauma Stress. 2005 Dec;18(6):607-16. doi: 10.1002/jts.20069. PMID 16382428
- [Background] Shapiro F, Maxfield L. Eye Movement Desensitization and Reprocessing (EMDR): information processing in the treatment of trauma. J Clin Psychol. 2002 Aug;58(8):933-46. doi: 10.1002/jclp.10068. PMID 12115716
- [Background] Striegel-Moore RH, Dohm FA, Pike KM, Wilfley DE, Fairburn CG. Abuse, bullying, and discrimination as risk factors for binge eating disorder. Am J Psychiatry. 2002 Nov;159(11):1902-7. doi: 10.1176/appi.ajp.159.11.1902. PMID 12411226
- [Background] Tagay S, Schlottbohm E, Reyes-Rodriguez ML, Repic N, Senf W. Eating disorders, trauma, PTSD, and psychosocial resources. Eat Disord. 2014;22(1):33-49. doi: 10.1080/10640266.2014.857517. PMID 24365526
- [Background] van der Kolk BA, Spinazzola J, Blaustein ME, Hopper JW, Hopper EK, Korn DL, Simpson WB. A randomized clinical trial of eye movement desensitization and reprocessing (EMDR), fluoxetine, and pill placebo in the treatment of posttraumatic stress disorder: treatment effects and long-term maintenance. J Clin Psychiatry. 2007 Jan;68(1):37-46. doi: 10.4088/jcp.v68n0105. PMID 17284128
- [Background] Wonderlich S, Mitchell JE. The role of personality in the onset of eating disorders and treatment implications. Psychiatr Clin North Am. 2001 Jun;24(2):249-58. doi: 10.1016/s0193-953x(05)70221-5. PMID 11416925
- [Background] Wonderlich SA, Mitchell JE. Eating disorders and comorbidity: empirical, conceptual, and clinical implications. Psychopharmacol Bull. 1997;33(3):381-90. PMID 9550882
- [Background] Wonderlich SA, Brewerton TD, Jocic Z, Dansky BS, Abbott DW. Relationship of childhood sexual abuse and eating disorders. J Am Acad Child Adolesc Psychiatry. 1997 Aug;36(8):1107-15. doi: 10.1097/00004583-199708000-00018. PMID 9256590
- [Background] Wonderlich SA, Crosby RD, Mitchell JE, Thompson KM, Redlin J, Demuth G, Smyth J, Haseltine B. Eating disturbance and sexual trauma in childhood and adulthood. Int J Eat Disord. 2001 Dec;30(4):401-12. doi: 10.1002/eat.1101. PMID 11746301